CLINICAL TRIAL: NCT05342194
Title: A Phase III, Randomized, Three-arm, Double-blind, Placebo-controlled, International Multi-center Study to Evaluate the Efficacy and Safety of Toripalimab in Combination With Lenvatinib and Gemcitabine-based Chemotherapy Compared With Gemcitabine-based Chemotherapy as First-line Treatment in Patients With Unresectable Advanced Intrahepatic Cholangiocarcinoma (ICC)
Brief Title: Toripalimab Plus Lenvatinib and Gemcitabine-based Chemotherapy in 1L Treatment of Advanced ICC: a Phase III Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JS001-039-III-ICC
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
Keywords: Intrahepatic cholangiocarcinoma; Toripalimab; lenvatinib; Chemotherapy
MeSH Terms: conditions — Cholangiocarcinoma | interventions — toripalimab; lenvatinib; Oxaliplatin; Injections; Gemcitabine; Cisplatin

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Toripalimab, lenvatinib, and gemcitabine-based chemotherapy-Arm A (Experimental): Toripalimab plus lenvatinib and GEMOX (Gemcitabine hydrochloride and Oxaliplatin for injection ) or GC (Gemcitabine hydrochloride and Cisplatin)
  Interventions: Drug: Toripalimab; Drug: Lenvatinib mesylate capsules; Drug: Oxaliplatin for injection; Drug: Gemcitabine hydrochloride; Drug: Cisplatin
- Toripalimab, oral placebo, and gemcitabine-based chemotherapy -Arm B (Experimental): Toripalimab plus lenvatinib placebo and GEMOX (Gemcitabine hydrochloride and Oxaliplatin for injection ) or GC (Gemcitabine hydrochloride and Cisplatin)
  Interventions: Drug: Toripalimab; Drug: Oral placebo; Drug: Oxaliplatin for injection; Drug: Gemcitabine hydrochloride; Drug: Cisplatin
- Intravenous placebo, oral placebo, and gemcitabine-based chemotherapy-Arm C (Active Comparator): Toripalimab placebo plus lenvatinib placebo and GEMOX (Gemcitabine hydrochloride and Oxaliplatin for injection ) or GC (Gemcitabine hydrochloride and Cisplatin)
  Interventions: Drug: Placebo IV; Drug: Oral placebo; Drug: Oxaliplatin for injection; Drug: Gemcitabine hydrochloride; Drug: Cisplatin

INTERVENTIONS:
Drug: Toripalimab — 240 mg IV on day 1 of each 21-day treatment cycle (Q3W) for up to 35 treatment cycles
  Other Names: Tuoyi
  Arms: Toripalimab, lenvatinib, and gemcitabine-based chemotherapy-Arm A; Toripalimab, oral placebo, and gemcitabine-based chemotherapy -Arm B
Drug: Lenvatinib mesylate capsules — 8 mg orally (po) once daily (QD)
  Other Names: LENVIMA
  Arms: Toripalimab, lenvatinib, and gemcitabine-based chemotherapy-Arm A
Drug: Placebo IV — Placebo IV on day 1 of each 21-day treatment cycle (Q3W) for up to 35 treatment cycles
  Other Names: Toripalimab placebo
  Arms: Intravenous placebo, oral placebo, and gemcitabine-based chemotherapy-Arm C
Drug: Oral placebo — Oral placebo po QD continuously
  Other Names: Lenvatinib mesylate capsules placebo
  Arms: Intravenous placebo, oral placebo, and gemcitabine-based chemotherapy-Arm C; Toripalimab, oral placebo, and gemcitabine-based chemotherapy -Arm B
Drug: Oxaliplatin for injection — 85 mg/m2 IV, on day 1 of each 21-day treatment cycle (Q3W) up to 8 cycles
Drug: Gemcitabine hydrochloride — 1 g/m2 IV, on day 1 and day8 of each 21-day treatment cycle (Q3W) up to 8 cycles
Drug: Cisplatin — 25 mg/m2 IV, on day 1 and day8 of each 21-day treatment cycle (Q3W) up to 8 cycles

SUMMARY:
This is a Phase III, prospective, randomized, three-arm, double-blind, placebo-controlled, international multicenter study to evaluate the efficacy and safety of toripalimab in combination with lenvatinib and gemcitabine-based chemotherapy compared with gemcitabine-based chemotherapy as first-line treatment for unresectable advanced ICC.

This study will enroll approximately 480 patients with unresectable advanced ICC who have received no prior systemic therapy. Patients who meet the requirements will be randomly assigned to Treatment Arm A: Toripalimab, lenvatinib, and gemcitabine-based chemotherapy or Treatment Arm B: Toripalimab, oral placebo, and gemcitabine-based chemotherapy or Treatment Arm C: Intravenous placebo, oral placebo, and gemcitabine-based chemotherapy.

All patients will receive standard chemotherapy (GEMOX or GC per Investigator decision) for a maximum of 8 cycles. After the completion of standard chemotherapy, all patients continue to receive maintenance therapy with toripalimab injection or its placebo in combination with lenvatinib mesylate capsule or its placebo until unacceptable toxicity, confirmed disease progression and loss of clinical benefit as determined by the investigators, start of new anti-cancer therapy, death, other conditions requiring termination of study treatment, or the patient meets the criteria for study withdrawal, whichever occurs first.

In the absence of unacceptable toxicity, patients who meet criteria for unconfirmed disease progression per RECIST v1.1 while receiving toripalimab, lenvatinib, or their placebos will be permitted to continue treatment if their clinical status or symptoms are stable or improved (as determined by the investigators) or until loss of clinical benefit. Patients with confirmed disease progression should discontinue toripalimab, lenvatinib, or their placebos.

Tumor assessments will be performed at screening and during the study treatment per protocol. In the absence of progression, tumor assessments will continue as scheduled, regardless of whether study treatment ends, until confirmed disease progression or other criteria for study withdrawal are met, whichever occurs first. Patients who meet RECIST v1.1 criteria for progression should undergo tumor assessments as scheduled if clinical benefits of continuing study treatment are determined by investigators until progression is confirmed per iRECIST (iCPD), or the criteria for study withdrawal are met, whichever occurs first.

Computerized tomography (CT)/magnetic resonance imaging (MRI) scans for efficacy evaluation will be performed at baseline, every 6 weeks (Q6W) in the first year (52 weeks), and every 9 weeks (Q9W) in the second year (after week 52).

All AEs and concomitant medications during the study will be recorded. An end-of-treatment (EOT) visit will be performed within 30 days after the last dose of study treatment or termination of study treatment is confirmed by the investigator. After the EOT visit, follow-up for survival (telephone visit is allowed) will be conducted and AEs and subsequent anti-cancer therapy will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18-75 years (inclusive), male or female;
2. Volunteer to participate in the study by signing the informed consent form and the ability to comply with the study protocol;
3. Advanced ICC with diagnosis confirmed by histology or cytology;
4. Stage II, III, or IV per TNM staging for ICC of the American Joint Committee on Cancer (AJCC) (8th edition, 2017). Those with Stage II or III should be determined to be unresectable by the investigator;
5. Patients with no prior systemic chemotherapy or targeted therapy or loco-regional therapy (including but not limited to transarterial chemoembolization, transarterial embolization, transarterial chemotherapy or transarterial radioembolization) for ICC. Patients with recurrent disease more than 6 months after completion of adjuvant chemotherapy following curative resection are eligible;
6. Measurable lesion per RECIST v1.1;
7. Child-Pugh class A with no history of hepatic encephalopathy;
8. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1;
9. Life expectancy ≥12 weeks;

Exclusion Criteria:

1. Diagnosis of hepatocellular carcinoma (HCC), mixed cholangiocarcinoma and HCC, sarcomatoid hepatocellular carcinoma, or hepatic fibrolamellar carcinoma by histology or cytology;
2. History of malignancy other than ICC within 5 years prior to screening, with the exception of localized malignancies that have been cured, including non-melanoma skin cancers, cervical carcinoma in situ, breast carcinoma in situ, and papillary thyroid carcinoma;
3. Prior radiotherapy for ICC within 4 weeks prior to randomization;
4. Major surgical procedures within 4 weeks prior to randomization;
5. Side effects from prior therapy (except alopecia and pigmentation) that has not recovered to ≤ grade 1 (per NCI-CTCAE v5.0) or levels specified in the inclusion/exclusion criteria;
6. Uncontrolled pericardial effusion, pleural effusion, or clinically significant moderate or severe ascites that is symptomatic or requires thoracentesis or paracentesis during the screening phase for control of symptoms;
7. Gastrointestinal (GI) hemorrhage within 6 months prior to randomization and/or gastrointestinal varices that have not been assessed and treated, if appropriate, within 6 months prior to randomization.
8. Gastrointestinal or non-gastrointestinal fistula, gastrointestinal perforation, or abdominal abscess within 6 months prior to randomization;
9. Ongoing or a history of recurrent intestinal obstruction. Patients with a single episode of intestinal obstruction that has fully resolved following treatment are eligible allowed;
10. History of serious cardiovascular and cerebrovascular diseases:
11. Significant bleeding and coagulopathy or other evidence of bleeding diathesis, to include:
12. Pre-existing CNS metastases and/or meningeal metastases (including dural metastases and leptomeningeal metastases);
13. Serious non-healing wound, active ulcer, or untreated bone fracture;
14. Vaccination with live virus or bacteria within 30 days prior to randomization;
15. Active autoimmune disease or history of autoimmune disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in Arm A compared with Arm C (OS A vs. C) | Until 2 years after the last subject was enrolled
  OS is defined as the time from randomization to death due to any cause. Overall survival will be compared between Arm A and Arm C

SECONDARY OUTCOMES:
OS in Arm B compared with Arm C (OS B vs. C) | Until 2 years after the last subject was enrolled
  OS is defined as the time from randomization to death due to any cause. Overall survival will be compared between Arm B and Arm C
Investigator-determined progression-free survival (PFS) | Until 2 years after the last subject was enrolled
  Investigator-determined progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (v1.1) in Arm A compared with Arm C (PFS A vs. C);
Investigator-determined progression-free survival (PFS) | Until 2 years after the last subject was enrolled
  Investigator-determined PFS according to RECIST v1.1 in Arm B compared with Arm C (PFS B vs. C);
Investigator-determined objective response rate (ORR) | Until 2 years after the last subject was enrolled
  Investigator-determined objective response rate (ORR) according to RECIST v1.1 in Arm A compared with Arm C (ORR A vs. C)
Investigator-determined objective response rate (ORR) | Until 2 years after the last subject was enrolled
  Investigator-determined ORR according to RECIST v1.1 in Arm B compared with Arm C (ORR B vs. C)

OTHER OUTCOMES:
OS rates | Until 2 years after the last subject was enrolled
  1-year and 2-year OS rates between Arm A and Arm C
OS rates | Until 2 years after the last subject was enrolled
  1-year and 2-year OS rates between Arm B and Arm C
adverse events (AE), immune-related adverse events (irAE) and serious adverse events (SAE) | Until 2 years after the last subject was enrolled
  To evaluate incidence, severity and outcome of adverse events (AE), immune-related adverse events (irAE) and serious adverse events (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No